CLINICAL TRIAL: NCT02346968
Title: Evaluation of Serum and Urinary C-terminal Agrin Fragment-22 (CAF22) as Novel Renal Function Marker in Kidney Transplant Recipients - A Prospective Observational Study
Brief Title: Evaluation of CAF22 After Renal Transplantation
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 98/14
Record Dates: First submitted 2015-01-20; First posted 2015-01-27 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Kidney Transplantation; Delayed Graft Function
Keywords: Kidney Transplantation; Delayed Graft Function; C-terminal fragment of agrin; Dialysis
MeSH Terms: conditions — Delayed Graft Function | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All study participants: Patients with end stage renal disease (ESRD) planned to undergo kidney transplantation.
  Interventions: Other: Blood and urine sampling

INTERVENTIONS:
Other: Blood and urine sampling — Blood and urine sampling (in the context of routine sampling)

SUMMARY:
Established markers of kidney function, such as creatinine, have considerable limitations in the diagnosis of delayed graft function (DGF) after kidney transplantation (KT). Indeed, creatinine does not accurately reflect minor changes of renal function as its levels change only upon significant fluctuations of the latter. CAF22 is a molecule which arises from the degradation of a larger protein and it is proposed to be a reliable and more sensitive marker of renal function. This study aims to further clarify this issue by measuring blood and urine concentrations of CAF22 and comparing them with creatinine levels before and after KT.

The main assumption is that blood CAF22 levels could serve as a more sensitive kidney function biomarker than creatinine post-KT to detect DGF.

DETAILED DESCRIPTION:
Background

Kidney transplantation (KT) is the most appropriate therapy of end stage renal disease (ESRD). While the number of kidney donors remained stable during the last decade the number of patients waiting for a kidney transplantation are rapidly increasing resulting in utilization of an increasing numbers of marginal renal transplants. These kidneys show a relatively high percentage of delayed graft function (DGF), which complicates post-transplant management and increases both the duration of initial hospitalization and the cost of transplantation.

Exact measurement of glomerular filtration rate (GFR) is complex in the clinical setting and thus GFR is usually estimated from serum creatinine levels through creatinine-based equations such as the MDRD or the CKD-EPI equations. Particularly, this is the case in kidney recipients with DGF, in whom creatinine levels remain high and they have to undergo dialysis. Creatinine is dialyzable, so that it cannot reflect the actual renal function in this setting due to fluctuations of its levels. Thus there is emergent need for a more accurate renal biomarker.

CAF22 is the C-terminal 22 kDa domain of agrin. Agrin is cleaved by its specific protease neurotrypsin at two distinct sites, whereas cleavage at the beta site generates a 22 kDa C-terminal fragment (CAF22). In the kidney agrin is part of the basal lamina, where it is the major contributor of the anionic potential of the glomerular basement membrane (GBM). There are indices for a proteolytic activity selectively shedding the C-terminal part of agrin of the GBM. Recently, a 19-fold increase of CAF22 levels in ESDR was observed, which was reduced in patients receiving KT, qualifying CAF22 as effective renal function marker. Additionally, current data support that CAF22 levels are not influenced by inflammatory processes, steroids or by hemodialysis with a standard dialysis membrane.

Objective

Primary:

- to compare CAF22 versus creatinine as biomarkers for DGF prediction in patients undergoing kidney transplantation

Secondary:

* to evaluate the kinetics of CAF levels related with the graft function outcomes "immediate graft function (IGF)" and "delayed graft function (DGF)"
* to elucidate whether CAF can make estimations on the required hemodialysis days of patients with delayed graft function

Methods

Research project with humans associated with the collection of biologic material and health-related data. Prospective, observational trial.

All patients will be screened consecutively before undergoing kidney transplantation (KT).

All participants will undergo blood and urine sampling for estimation of CAF22 levels once before KT, once daily during the first 7 days after KT as well as at 2, 4 and 12 weeks after KT. Blood and urine sampling for CAF22 will be performed during routine follow-up sampling.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Written informed consent
* All patients planned to undergo kidney transplantation

Exclusion Criteria

* Age <18 years old
* Pregnancy
* Other individuals especially in need of protection (according to the Swiss Academy of Medical Sciences)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with end stage renal disease (ESRD) planned to undergo kindey transplantation in Bern University Hospital will be screened consecutively, informed and asked for written inform consent.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2014-10-08 (Actual); Primary Completion 2018-09-27 (Actual); Study Completion 2018-09-27 (Actual)

PRIMARY OUTCOMES:
Delayed graft function (DGF) defined as the requirement of dialysis within 7 days after transplantation | 7 days

SECONDARY OUTCOMES:
Immediate graft function (IGF) | 7 days
Need for hemodialysis | 7 days
Hemodialysis duration (in days) | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Spyridon Arampatzis, MD, Principal Investigator — Dep. of Nephrology, Hypertension and Clinical Pharmacology, Bern University Hospital, Bern, Switzerland
Locations (2):
- Department of Nephrology, University Hospital of Essen, Essen, Germany
- Dep. of Nephrology, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Steubl D, Hettwer S, Vrijbloed W, Dahinden P, Wolf P, Luppa P, Wagner CA, Renders L, Heemann U, Roos M. C-terminal agrin fragment--a new fast biomarker for kidney function in renal transplant recipients. Am J Nephrol. 2013;38(6):501-8. doi: 10.1159/000356969. Epub 2013 Dec 14. PMID 24356308
- [Background] Steubl D, Hettwer S, Dahinden P, Wolf P, Luppa P, Wagner CA, Kuchle C, Schmaderer C, Renders L, Heemann U, Roos M. Influence of high-flux hemodialysis and hemodiafiltration on serum C-terminal agrin fragment levels in end-stage renal disease patients. Transl Res. 2014 Nov;164(5):392-9. doi: 10.1016/j.trsl.2014.05.005. Epub 2014 May 16. PMID 24907476
- [Background] Steubl D, Hettwer S, Dahinden P, Luppa P, Rondak IC, Regenbogen C, Stock KF, Renders L, Heemann U, Roos M. C-terminal agrin fragment (CAF) as a serum biomarker for residual renal function in peritoneal dialysis patients. Int Urol Nephrol. 2015 Feb;47(2):391-6. doi: 10.1007/s11255-014-0852-5. Epub 2014 Oct 29. PMID 25352149
- [Background] Ojo AO, Wolfe RA, Held PJ, Port FK, Schmouder RL. Delayed graft function: risk factors and implications for renal allograft survival. Transplantation. 1997 Apr 15;63(7):968-74. doi: 10.1097/00007890-199704150-00011. PMID 9112349
- [Background] Levey AS, Stevens LA, Schmid CH, Zhang YL, Castro AF 3rd, Feldman HI, Kusek JW, Eggers P, Van Lente F, Greene T, Coresh J; CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration). A new equation to estimate glomerular filtration rate. Ann Intern Med. 2009 May 5;150(9):604-12. doi: 10.7326/0003-4819-150-9-200905050-00006. PMID 19414839